CLINICAL TRIAL: NCT05829824
Title: Connect Cancer Patients to Tobacco Cessation Care by Automated Interactive Outreach
Brief Title: Tobacco Cessation Care for Cancer Patients by Automated Interactive Outreach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 226310; NCI-2023-03215 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Tobacco Dependence; Tobacco Use Cessation
Keywords: Interactive Intervention
MeSH Terms: conditions — Neoplasms; Tobacco Use Disorder; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CareConnect (Intervention) (Experimental): Participants will receive automated 'CareConnect' calls/SMS text at enrollment. The call protocol includes up to 2 calls on 2 consecutive days if no response to first call. If there is no response to call, a follow up SMS 3-4 days later. Each CareConnect contact will include (1) assessment, (2) motivational enhancement tailored to participants' tobacco use status and importance of quitting; and (3) multiple referral options (UCSF Fontana Tobacco Treatment Center (FTTC)/tobacco treatment specialist, Quitline, or smoke-freeTXT from smokefree.gov), offered after the motivational enhancement message. CareConnect will notify UCSF tobacco treatment specialist of participants acceptance of any of referral options. Referral options will be documented by specialists on the participants electronic health record (EHR). Participants who have completed the CareConnect call will be contacted by research staff for a 3-month survey to be completed online, by telephone, or postal mail.
  Interventions: Behavioral: CareConnect; Procedure: Biospecimen samples
- AutoReach (Control) (Other): Participants will receive automated AutoReach calls/Short Message Service (SMS) text at enrollment provides one referral option (speaking with a tobacco treatment specialist) and an option for sending information on cessation resources. All participants who have completed the AutoReach call will be contacted by research staff for a 3-month survey to be completed online, by telephone or postal mail.
  Interventions: Other: AutoReach; Procedure: Biospecimen samples

INTERVENTIONS:
Behavioral: CareConnect — A combination of the Ask-Advise-Connect (AAC) with an Interactive Voice Response (IVR)
  Other Names: Automated Interactive Outreach
  Arms: CareConnect (Intervention)
Other: AutoReach — Phone call / SMS Text
  Other Names: Automated Interactive Outreach
  Arms: AutoReach (Control)
Procedure: Biospecimen samples — Optional saliva sample
  Other Names: Biological Specimens

SUMMARY:
This is a multi-arm, randomized controlled, pilot study which will recruit cancer patients who have been seen by a UCSF Cancer Center-affiliated clinical department to evaluate the efficacy of "CareConnect". This is the first study to assess the efficacy CareConnect, a combination of the Ask-Advise-Connect (AAC) with an Interactive Voice Response (IVR) delivering cancer-targeted educational messages to support referral to smoking cessation resources for patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate CareConnect's efficacy on referring patients to tobacco cessation resources.

SECONDARY OBJECTIVE:

I. To evaluate patients' acceptance of referrals.

II. To evaluate the acceptability of CareConnect.

EXPLORATORY OBJECTIVES:

I. In-depth semi-structured qualitative interviews of 20 selectively chosen participants who completed the 3-month follow-up survey or finished the automated CareConnect or Auto-Reach call but may have refused to complete the 3-month follow-up survey (10 from each group).

II. Smoking cessation with verification.

OUTLINE:

Eligible participants, identified through the Cancer Center Tobacco Registry will be randomized to either the Intervention or Control arm on a 1:1 ratio. Participants who complete the first call of CareConnect or AutoReach will be considered enrolled. Participants will complete a baseline assessment, a 3-month assessment, and have option to provide a saliva sample.

For those who are selected to participate in an in-depth interview, this will take place within 1 month after the 3-month assessment. Data from the participants medical record may be accessed at 6 months post follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older.
2. Able to understand study procedures and to comply with them for the entire length of the study.
3. Ability of individual or legal guardian/representative to understand a written informed consent document, and the willingness to sign it.
4. English, Spanish, Cantonese, or Mandarin speaking.
5. Self-reported current use of tobacco, including e-cigarette on EHR.
6. Has a diagnosis of cancer.
7. Has been seen by a prescribing provider within a UCSF Cancer Center-affiliated clinical department within the past 3 months.

Exclusion Criteria:

1. Contraindication to any study-related procedure or assessment.
2. No valid contact telephone number.
3. Currently hospitalized or having been discharged from inpatient setting within the past month (according to EHR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who report using any smoking cessation resources | Up to 3 months
  Self-reported receipts (recorded as 'yes' or 'no') of evidence-based, smoking cessation services assessed at 3 months post-intervention will be reported as a proportion.

SECONDARY OUTCOMES:
Proportion of participants who started the call and chose the referrals | Up to 3 months
  Proportion of participants who started the call and chose the referrals to quitline/speaking with a tobacco treatment specialist or to use smokefree.gov
Mean Satisfaction Ratings (CareConnect Group Only) | Up to 3 months
  Participants in the CareConnect intervention group will be asked to respond to the following single item to measure overall satisfaction with the CareConnect intervention from answers to the following question "How helpful was the call you received about tobacco use and cancer care?". The response to this single item is scored on a range from 0= 'Not at all helpful' to 4= 'Extremely helpful'. Higher scores indicate a greater degree of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No